CLINICAL TRIAL: NCT02167165
Title: Role of Genetic Factors in the Response to Digoxin in the Acute Treatment of Atrial Fibrillation
Brief Title: Role of SNP and DIGOXIN Response in Atrial Fibrillation Patients
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Other Study IDs: AF/DIGOXIN
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Digoxin; SNP
MeSH Terms: conditions — Atrial Fibrillation | interventions — Digoxin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — arterial blood samples collected in EDTA tubes and stored in - 20°C envirement for DNA extraction with salting out methods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Digoxin and AF: Patients consulting the emergency deprtment (ED) for AF and receiving Digoxin treatment
  Interventions: Drug: Digoxin Injection

INTERVENTIONS:
Drug: Digoxin Injection — Patients consulting the ED for Acute onset AF received 0.5 mg digoxin by oral root

SUMMARY:
This study tested the hypothesis that response to digoxin is modulated by single Nucleotid Polymorphism (SNP):

* Multi Drug Resistance (MDR1) gene haplotypes and Solute carrier organic anion transporter family member 1B3 (SLCO1B3) gene Polymorphism and their role in the response to treatement.
* Aldosterone synthase (CYP11B2) gene and sodium channel, voltage-gated, type V alpha subunit gene (SCN5A) correlated with atrial fibrillation and their roles in response to digoxin.

DETAILED DESCRIPTION:
The frequency distribution of single nucleotide polymorphisms (SNPs) and haplotypes in the ABCB1 and SLCO1B3 genes varies largely among populations. The aim of this study is to investigate the genomic variations influence of these two genes on the response to digoxin in Tunisian atrial fibrillation (AF) patients.

In fact human P-glycoprotein (P-gp) is encoded by the ABCB1 gene (MDR1), which is located on chromosomal region 7q21 and consists of 28 exons. To date, over 50 SNPs have been reported for this gene, some of them are known to be of functional relevance and can also alter the pharmacokinetics of substrate drugs. The aim of the current study is to analyze the ABCB1: C1236T (Gly412Gly), G2677>T⁄A (Ala893Ser/ Thr) and C3435T (Il1145Ile) polymorphisms.

SLCO1B3 (OATP1B3) gene located on chromosomal region 12p12 is highly polymorphic. It is known to transport digoxin and expressed on the sinusoidal membranes of hepatocytes in humans. It mediated uptake into hepatocytes and may be an important step of the elimination of digoxin. In this study we will also investigate the relationship between two deletion polymorphisms (from -28 to -11 deletion) and (from-7 to -4 deletion), T334G (Ser112Ala) and G699A (Met233Ile) SNPs in the SLCO1B3gene and their role in response to digoxin.

Another way, progress in understanding molecular mechanisms in AF supports the idea that variability in response to drug therapy may reflect differences in disease mechanisms, it is entirely possible that response to AF is highly heterogeneous because the arrhythmia itself is not a single pathophysiologic entity.

Aldosterone synthase (CYP11B2) gene polymorphism was found to be correlated with atrial fibrillation (AF) risk. Moreover, the human cardiac sodium channel SCN5A is responsible for the fast depolarization upstroke of the cardiac action potential and serves as a molecular target for antiarrhythmic drugs. Mutations in the human cardiac sodium channel gene have been previously discovered in a spectrum of cardiac rhythm disorders. We hypothesized that the T-344C and H558R (His558Arg) SNPs in CYP11B2 and SCN5A gene which are associated with susceptibility to AF could be implicated in the variation of response to Digoxin.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 20 years
* Quick AF (heart rate> 120 bpm) diagnosed by ECG

Exclusion Criteria:

* HR under 120 bpm
* Hemodynamically unstable patients
* Atrio-Ventricular-block (second or third degree)
* Ventricular rhythm disorder
* Acute coronary syndrome
* kidney failure
* Hypokalimia

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting at the ED with acute onset AF documented by ECG.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Correlation between the response to digoxin and the genotypes of the patients | 24 hours
  In the current study we aimed at outlining the different MDR-1, SLCO1B3, CYP11B12 and SCN5A genotypes in a sample of Tunisian patients, suffering from AF and taking digoxin, to assess the role of SNPs in affecting serum digoxin concentrations, and studying the consequences on patients' clinical outcome. Patients will be monitored for 24 hours in an intensive care unit;

SECONDARY OUTCOMES:
Rhythm and Rate control | 24 hours
  Rhythm control: rate and delay of return to sinusal rhythm. Rate control: reduction of heart rate : HR <100 bpm or 20% reduction from baseline

OTHER OUTCOMES:
Arterial hypotension Bradycardia (HR <45 bpm) Other (chest pain, allergic reaction……) | 24 hours
  hypotension during hospitalisation, bradycardia, chest pain, allergic reaction

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Samir, Professor, Principal Investigator — University of Monastir
Locations (1):
- university of Monastir, Monastir, Tunisia

REFERENCES:
- See also: official website — http://www.urgencemonastir.com